CLINICAL TRIAL: NCT03334877
Title: Cervicovaginal Fluid B-hCG Versus Fetal Fibronectin Assay in Prediction of Preterm Labor in Asymptomatic High Risk Women
Brief Title: Prediction of Preterm Labor in Asymptomatic High Risk Women
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed lotfy, assistant Professor of Obstetrics and Gynecology, Zagazig University
Other Study IDs: ZUH 50
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- β -human chorionic gonadotropin: Cervico vaginal fluid sampling was undertaken for qualitative assessment of β -human chorionic gonadotropin (β-hCG) and fetal fibronectin(fFN) at 24 weeks of gestation to predict preterm labour in asymptomatic high risk patients
  Interventions: Diagnostic Test: β -human chorionic gonadotropin

INTERVENTIONS:
Diagnostic Test: β -human chorionic gonadotropin — Cervico vaginal fluid sampling was undertaken for qualitative assessment of β -human chorionic gonadotropin (β-hCG) and fetal fibronectin(fFN) at 24 weeks of gestation.

SUMMARY:
Two hundred and twenty women with singleton pregnancies and risk factors for spontaneous preterm birth were included in this study. Cervico vaginal fluid sampling was undertaken for qualitative assessment of β -human chorionic gonadotropin (β-hCG) and fetal fibronectin(fFN)at 24 weeks of gestation.

For qualitative assay of both b-hCG and fFN, first vaginal specimens were collected by the following method:

Specimen collection

A sterile Cusco speculum was introduced into the vagina; the anterior lip of the cervix was grasped with sponge forceps and a cotton-tipped swab was placed into the external part of the endocervical canal (not reaching the internal os) and then into the posterior fornix (each for at least 1 min) to obtain an adequate sample of cervico vaginal secretions. Sampling was performed before doing any cervical manipulation (digital or ultrasound examination) and before introducing any vaginal material (lubricants or medications). The Hologic Specimen Collection Kit is the only acceptable specimen collection system which can be used to collect specimens for this assay. The polyester tipped swab provided in the Specimen Collection Kit should be inserted into the vagina and lightly rotated across the posterior fornix for approximately 10 seconds to absorb the cervico vaginal secretions. Once the specimen is obtained, carefully remove the swab from the vagina and place it into the tube of buffer provided with the Specimen Collection Kit. Two Specimen Collection Device per patient were obtained; one for each assay. Label the Specimen Transport Tubes with the patient's name and any other identifying information required.

All women were then followed up till delivery. Women were categorized into two arms: women who delivered preterm (before 37 completed weeks of gestation) and women who delivered at term (after 37 completed weeks of gestation).

DETAILED DESCRIPTION:
Patients and methods

This prospective observational study was undertaken from May 2015to October 2017 at Zagazig university hospitals.This study was approved by the Research Ethical Committee of Zagazig university hospital. Written informed consent was obtained from all participants. Two hundred and twenty women with singleton pregnancies and risk factors for spontaneous preterm birth were included in this study. Cervico vaginal fluid sampling was undertaken for qualitative assessment of β -human chorionic gonadotropin (β-hCG) and fetal fibronectin (fFN) at 24 weeks of gestation.

Inclusion criteria:

There were past history of one or more spontaneous preterm labor or preterm rupture of membranes at less than 37 weeks of gestation, previous spontaneous second trimester miscarriage, previous cervical surgery (large loop excision of the transformation zone, loop electro surgical excision procedure, laser or cone excision), or an accidental finding of a cervical length of 25 mm or less in the current pregnancy.

Exclusion criteria:

Women who reported prior sexual intercourse (within 24 hours), or confirmed or suspected rupture of membranes, or who had vaginal bleeding visible on the swab.

Gestational age was confirmed by early obstetric ultrasonography (11-14 weeks of gestation). Participant baseline demographic data, obstetric history, and risk factors were tabulated and analysed.

For qualitative assay of both b-hCG and fFN, first vaginal specimens were collected by the following method:

Specimen collection

A sterile Cusco speculum was introduced into the vagina; the anterior lip of the cervix was grasped with sponge forceps and a cotton-tipped swab was placed into the external part of the endocervical canal (not reaching the internal os) and then into the posterior fornix (each for at least 1 min) to obtain an adequate sample of cervico vaginal secretions. Sampling was performed before doing any cervical manipulation (digital or ultrasound examination) and before introducing any vaginal material (lubricants or medications). The Hologic Specimen Collection Kit is the only acceptable specimen collection system which can be used to collect specimens for this assay. The polyester tipped swab provided in the Specimen Collection Kit should be inserted into the vagina and lightly rotated across the posterior fornix for approximately 10 seconds to absorb the cervico vaginal secretions. Once the specimen is obtained, carefully remove the swab from the vagina and place it into the tube of buffer provided with the Specimen Collection Kit. Two Specimen Collection Device per patient were obtained; one for each assay. Label the Specimen Transport Tubes with the patient's name and any other identifying information required.

Qualitative assessment of β-hCG assessment

The qualitative assay of β-hCGwas performed as a bedside test. The swab was then inserted in a tube containing 0.75 ml of sterile normal saline for dilution. From this sample, three drops were used for a bedside HCG test using ACON-HCG one-step pregnancy test strip (Rapid diagnostic Pvt. Ltd, India). with a detection cut-off value of 25 mIU/ ML.

Qualitative assessment of fFNtest:

It was done using Quick Check fFN test; it is a 10-minute, one-step, visual test. The test strip was removed from the foil pouch and its lower end (indicated by the arrows) was inserted into the tube containing the extraction buffer for 10 minutes. A positive sample contain fFN will result in two lines in test strip and a negative sample will result in one control line in test strip.

All women were then followed up till delivery. Women were categorized into two arms: women who delivered preterm (before 37 completed weeks of gestation) and women who delivered at term (after 37 completed weeks of gestation).

Those women who had iatrogenic preterm labor due to fetal or maternal indications were excluded from the final statistical analysis and were calculated among the women who did not complete follow up. Only women with spontaneous preterm labor were included.

Pregnancy outcome details were obtained from handheld notes, reviewed by trained research midwives, and entered onto the study database. Data entry was checked for inaccuracies contemporaneously by senior research midwives. Women were considered to have the outcome of interest (spontaneous preterm birth) if they had spontaneous onset of labor, or experienced preterm premature rupture of membranes with subsequent premature delivery

ELIGIBILITY:
Inclusion Criteria:

* There were past history of one or more spontaneous preterm labor or preterm rupture of membranes at less than 37 weeks of gestation.
* previous spontaneous second trimester miscarriage.
* previous cervical surgery (large loop excision of the transformation zone, loop electrosurgical excision procedure, laser or cone excision).
* accidental finding of a cervical length of 25 mm or less in the current pregnancy.

Exclusion Criteria:

* Women who reported prior sexual intercourse (within 24 hours).
* confirmed or suspected rupture of membranes.
* vaginal bleeding visible on the swab.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Two hundred and twenty women with singleton pregnancies and risk factors for spontaneous preterm birth were included in this study at 24 weeks of gestation.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
The diagnostic accuracy of qualitative level of cervico vaginal β-hCG versus fetal fibronectin | From 24 weeks gestation till delivery
  Prediction of preterm labor in asymptomatic high risk women during antenatal care.